CLINICAL TRIAL: NCT03168646
Title: Comparative Study Between Arthroscopic Wafer and Ulnar Shortening Osteotomy in Ulnar Abutment Syndrome
Brief Title: Arthroscopic Wafer and Ulnar Shortening in Ulnar Abutment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abd Elaziz Monsef Ali, principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WAFER
Record Dates: First submitted 2017-05-16; First posted 2017-05-30 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Wrist Impaction
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): wafer group procedure using an arthroscope through portal(radial to extensor carpi ulnaris, debridement of triangular fibro-cartilage complex 3-4 mm is shaved from the dome of the ulna by 2.9 bur.
  Interventions: Procedure: wafer procedure
- group 2 (Active Comparator): ulnar shortening group :this is the most logical technique, dorsoulnar incision is made on the distal one-third of the forearm then a 6 hole 3.5 mm Dcp plate is position,osteotomy using oscillating saw in z-shaped manner.
  Interventions: Procedure: arthroscopy and ulnar shortening osteotomy

INTERVENTIONS:
Procedure: wafer procedure — wrist arthroscopy and debridement of Triangular fibrocartilage and shortening of the head ulna by burr
  Arms: group 1
Procedure: arthroscopy and ulnar shortening osteotomy — wrist arthroscopy,debride debridement of Triangular fibrocartilage and shortening of the ulna by osteotomy and plate
  Arms: group 2

SUMMARY:
there are many management options of ulnocarpal abutment depends on clinical evaluation and imaging of this joint. Arthroscopic treatment is the simplest solution for these conditions.

ELIGIBILITY:
Inclusion Criteria:

* obvious ulnar abutment syndrome with ulnar side wrist pain

Exclusion Criteria:

* ulnar minus or neutral variance
* central and radial wrist pain
* osteoarthritis of the wrist.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
mayo scoring system | 6 month
  follow up of the pain( nonpain,mild occasional, moderate and sever graded as 1,2,3,4 respectively
mayo scoring system | 6 month
  Range of motion of the wrist compared to the normal side(100 ,75-99,50-74,25-9,0-24%
mayo scoring system | 6 month
  grip strength

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stockton DJ, Pelletier ME, Pike JM. Operative treatment of ulnar impaction syndrome: a systematic review. J Hand Surg Eur Vol. 2015 Jun;40(5):470-6. doi: 10.1177/1753193414541749. Epub 2014 Jul 30. PMID 25080480
- [Background] Kaufman D, Etcheson J, Yao J. Microfracture for Ulnar Impaction Syndrome: Surgical Technique and Outcomes with Minimum 2-Year Follow-up. J Wrist Surg. 2017 Feb;6(1):60-64. doi: 10.1055/s-0036-1586496. Epub 2016 Aug 5. PMID 28119797
- [Background] Colantoni J, Chadderdon C, Gaston RG. Arthroscopic wafer procedure for ulnar impaction syndrome. Arthrosc Tech. 2014 Jan 24;3(1):e123-5. doi: 10.1016/j.eats.2013.09.008. eCollection 2014 Feb. PMID 24749031